CLINICAL TRIAL: NCT00649415
Title: A Double Blind, Double Dummy, Randomized, Comparative Study Of The Efficacy And Safety Of Valdecoxib 40 Mg BID, PRN In The First Menstrual Cycle Day And Then Once A Day, And Piroxicam 40 Mg Once A Day In The Treatment Of Patients With Primary Dysmenorrhea
Brief Title: A Double Blind, Double Dummy, Randomized, Comparative Study Of The Efficacy And Safety Of Valdecoxib 40 Mg Twice Daily, As Needed In The First Menstrual Cycle Day And Then Once A Day, And Piroxicam 40 Mg Once A Day In The Treatment Of Patients With Primary Dysmenorrhea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: VALA-0513-137; A3471081
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea | interventions — Piroxicam; valdecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Drug: piroxicam
- Arm 2 (Active Comparator)
  Interventions: Drug: valdecoxib

INTERVENTIONS:
Drug: piroxicam — piroxicam 40 mg capsule QD for up to the first 3 days of the menstrual cycle
  Arms: Arm 1
Drug: valdecoxib — valdecoxib 40 mg capsule twice a day (BID), taken as required, on the first day of treatment in the menstrual cycle followed by oral valdecoxib 40 mg once a day (QD) for up to the first 3 days of the menstural cycle
  Arms: Arm 2

SUMMARY:
To compare the analgesic efficacy, safety, and tolerability of valdecoxib versus piroxicam in subjects with moderate to severe menstrual cramping pain associated with primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* History of primary dysmenorrhea with moderate to severe menstrual cramping pain for which the patient took analgesic medication for at least three of six previous menstrual cycles before enrollment
* Subjects were to have been in good health and were to have had a complete physical exam (including a pap smear and an endovaginal or pelvic ultrasound, unless the subject had had these examinations performed within 6 months prior to the Screening Visit and the results were normal) prior to inclusion

Exclusion Criteria:

* Subjects who were pregnant, lactating, breastfeeding or not using adequate methods of birth control

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2003-01; Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Total pain relief were calculated as the summed weighted pain releif scores | 8 hours

SECONDARY OUTCOMES:
adverse events | approximately 5 days after treated cycle
laboratory analyses | screening
Subjects' global evaluation of the study drug | 8 hours and 72 hours
Summed pain intensity difference | 8 hours
Percent of subjects who took rescue medication | 72 hours
Percent of subjects who took the second dose of study medication | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- Brazil (7):
  - Pfizer Investigational Site, Salvador, Estado de Bahia
  - Pfizer Investigational Site, Goiânia, Goiás
  - Pfizer Investigational Site, Belo Horizonte, Minas Gerais
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, São Paulo, São Paulo
  - Pfizer Investigational Site, São Paulo

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=VALA-0513-137